CLINICAL TRIAL: NCT06586385
Title: The Effect of ADDIE Model Based Training Given to Women on General Disaster Preparedness Belief Level and Disaster Literacy
Brief Title: The Effect of Education Given to Women on General Disaster Preparedness Belief Level and Disaster Literacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Selen ÖZDEMİR, Ataturk University, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Selen_Doktora_Tezi
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Disaster Education
Keywords: ADDIE Model; Disaster Literacy,; General Disaster Preparedness Belief Level; Nursing

STUDY DESIGN:
Intervention Model Description: The simple random sampling method will be used among the women who took the handicraft technology course at Erzincan Public Education Center, which constitutes the sample of the research. According to the sample pool formed by the women included in the research, the participants will be assigned to 2 groups as experimental and control with the "Research Randomizer" program (https://www.randomizer.org/). Each group will consist of at least 60 people.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The sample will consist of 30 women who are taking a course in the field of handicraft technology at the Public Education Center affiliated to the Erzincan Provincial Directorate of National Education and who are assigned through simple randomization to meet the conditions for inclusion in the study and who voluntarily consent to participate.
  Interventions: Behavioral: disaster education
- Control group (No Intervention): The sample will consist of 30 women who are taking a course in the field of handicraft technology at the Public Education Center affiliated to the Erzincan Provincial Directorate of National Education and who are assigned through simple randomization to meet the conditions for inclusion in the study and who voluntarily consent to participate.

INTERVENTIONS:
Behavioral: disaster education — The ADDIE Instructional Design Model will be used due to its suitability for adult education. General Disaster Awareness Training will be prepared according to the ADDIE instructional design model, which consists of five stages: analysis, design, development, implementation and evaluation. The trainings to be given will be given 1 week after the pre-test, 1 training per week, for a total of 3 trainings.
  Arms: Experimental group

SUMMARY:
It is aimed to determine the effect of the ADDIE Model-based training given to women on the level of disaster awareness and disaster literacy and to present suggestions for situations where deficiencies are observed based on the findings obtained.

DETAILED DESCRIPTION:
This research is a randomized controlled pre-test post-test experimental study aiming to evaluate the effect of the training to be provided. The research data is planned to be collected from women aged 18-60 who voluntarily agreed to participate in the research by taking a handicraft technology course at the Public Education Center affiliated to the Erzincan Provincial Directorate of National Education between April 2024 - April 2025.

The research universe will consist of women who took a handicraft technology course at the Public Education Center affiliated to the Erzincan Provincial Directorate of National Education between the data collection dates, and the sample will consist of 60 women who meet the conditions for inclusion in the research and who voluntarily consent to participate. The individuals constituting the sample will be divided into 2 equal groups by simple randomization.

Sample size of the research; The sample size for the research was determined by power analysis. In the power analysis, it was determined that a total of 52 people should be reached to reach 80% power at a 95% confidence interval at a significance level of 0.05 and a significance level of p<0.05. Considering that there may be data losses in the study, it was decided to reach 15% more of the sample, 60 people (30 experimental, 30 control) (Çapık, 2014).

All questions in the data collection tools (Personal Information Form, Disaster Literacy Scale, General Disaster Preparedness Belief Scale) will be transferred by the researchers and a form will be created for the pre-test. The created form will be applied face to face by the researchers to women who meet the criteria for inclusion in the study and they will be asked to answer all the questions completely.

After the collection of pre-test data in women in our study; It includes the training program to be given to the experimental group based on the ADDIE Model and the post-test to be applied to both groups. The ADDIE Instructional Design Model will be used in this study due to its suitability for adult education. General Disaster Awareness Training will be prepared according to the ADDIE instructional design model consisting of five stages: analysis, design, development, implementation and evaluation. The trainings to be given will be given 3 times in total, 1 training per week, 1 week after the pre-test.

The researchers will not make any interventions to the control group during this period. After the post-test is applied, the educational materials given to the experimental group will be given to the women in the control group.

After the training is completed, all the questions in the data collection tools (Personal Information Form, Disaster Literacy Scale, General Disaster Preparedness Belief Scale) will be transferred by the researchers and a form will be created for the post-test. One week after the training is completed, both groups will be asked to answer all the questions in the created form completely.

From this perspective, it is thought that this research will contribute to the development and dissemination of similar programs by increasing disaster literacy by replacing women's negative beliefs about general disaster preparedness with positive beliefs through the ADDIE Model-based training given to women.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-60,
* Being female,
* Agreeing to participate in the research,
* Not having a mental illness,
* Being literate and accessible,
* Not having a communication barrier,
* Not having received any training on disaster awareness, preparation before, during and after the disaster, and first aid in disasters.

Exclusion Criteria:

* Having received pre-disaster preparation training,
* Having received disaster management training,
* Having received post-disaster intervention training,
* Having received disaster first aid training,
* Women who are not between the ages of 18-60,
* Having a communication barrier,
* Having a mental illness

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Being between the ages of 18-60, not having a mental illness, being literate, accessible, and having no communication barriers.
Enrollment: 60 (Estimated)
Dates: Start 2024-09-03 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-04-18 (Estimated)

PRIMARY OUTCOMES:
The education given to women based on the ADDIE Model positively affects the general disaster preparedness belief level. | 1 week before the education and 1 week after the education
  İn order to assess the general disaster preparedness belief level of women, the General Disaster Preparedness Belief Scale will be administered 1 week before and 1 week after the ADDIE Model-based education.
The education given to women based on the ADDIE Model positively affects the level of disaster literacy. | 1 week before the education and 1 week after the education
  İn order to assess the disaster literacy level of women, the Disaster Literacy Scale will be administered 1 week before and 1 week after the ADDIE Model-based education.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk, Zubeyde Hanim St. No: 10, 24180 Erzincan Center/Erzincan, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No